CLINICAL TRIAL: NCT06029556
Title: Effects of Early Mobilization on Functional Capacity, Physical Activity and Kinesiophobia in Post Coronary Artery Bypass Grafting
Brief Title: Effects of Early Mobility Protocols in Cardiac ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REC/01373 Sarmad
Record Dates: First submitted 2022-12-06; First posted 2023-09-08 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: CABG
Keywords: Early mobility; Physical activity; Kinesiophobia; Functional capacity
MeSH Terms: conditions — Motor Activity; Kinesiophobia | interventions — Ergometry; Beds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobility out of Bed (Active Comparator)
  Interventions: Other: Mobility out of Bed; Other: Ergometry in Bed
- Ergometry in Bed (Experimental)
  Interventions: Other: Mobility out of Bed; Other: Ergometry in Bed

INTERVENTIONS:
Other: Mobility out of Bed — Active upper limb exercises will be conducted (flexion-extension and adduction-abduction) of large joints (shoulder, elbow and wrist) Associated with upper limb exercises, patients will undergo a series of exercises ergometer with lower limb (LL). The mobilization will be conduct on a cycle ergometer in an active, lasting 20 minutes, divided into three steps: heat 5 minutes; 10 minutes of low-intensity exercise, with a speed of 30 revolutions per minute (rpm); and 5 minutes recovery. The patient remains in the supine position with the head of the bed elevated to 45 degrees, while the lower limbs will remain planned
Other: Ergometry in Bed — Ankle pumps (5*2), knee extension (5*2), breathing exercises with elbow flexion and extension(5*2), spirometry and progressive early ambulation (from bed to wheelchair and wheelchair to standing and from standing to few steps), and conventional chest physical activity (5 minutes on precursor)

SUMMARY:
In this study the investigator aim to find the effects of early mobility on different physical activity protocols in post CABG patients. Physical activity, functional status, functional capacity, Kinesiophobia, ICU mortality, heart rate, blood pressure, oxygen saturation, length of hospital stay and sternal instability. To compare the physical activity protocol used by physical therapist.

DETAILED DESCRIPTION:
Current study will compare two different early mobility protocols and will help in assessing best protocol to be use in cardiac ICU for better outcomes of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Both Genders
* Extubated patients with no Complication
* Post CABG (Elective)
* Vitally stable
* 1st CABG
* Selective CABG surgeries

Exclusion Criteria:

* Post anesthesia Psychosis
* Corrective surgeries
* Post CABG Stroke
* Infectious wound
* Participants with a physical disability
* Intra-aortic balloon pump (IABP)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Functional Status score Questionnaire | Pre Operative (Baseline), 1st Assessment (0 Week) and 2nd Assessment (4 week)
  Five item scale measures the physical performance of patients in ICU.The Functional Status Score for the Intensive Care Unit (FSS-ICU) is a 5-item performance-based measure that utilizes an 8 point, ordinal scale to measure physical function for patients in the intensive care unit setting.
BAECK PHYSICAL ACTIVITY QUESTIONNAIRE | Pre Operative (Baseline), 1st Assessment (0 Week) and 2nd Assessment (4 week)
  Evaluates the physical activity over the past 12 months. The MBPAQ (BHPAQ) evaluates habitual physical activities in individuals. Activities are scored on a scale of 1-5. A score of 5 indicates the most activity and 1 indicates the least activity for each index.
6 minute walk Test | Pre Operative (Baseline), 1st Assessment (0 Week) and 2nd Assessment (4 week)
  Sub-maximal test evaluates the aerobic endurance. The 6-minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
Tampa Scale of Kinesiophobia | Pre Operative (Baseline), 1st Assessment (0 Week) and 2nd Assessment (4 week)
  Evaluate the fear of movement during activity ,17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. Individual item scores range from 1-4, with the negatively worded items (4,8,12,16) having a reverse scoring (4-1). The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia. Changes will be measured at baseline and at completion of 4th week

SECONDARY OUTCOMES:
STERNAL INSTABILITY SCALE: | Pre Operative (Baseline), 1st Assessment (0 Week) and 2nd Assessment (4 week)
  The sternal instability scale (SIS) is a non-invasive manual assessment tool used to detect early bony non-union or instability.
BORG RATING OF PERCEIVED EXERTION | Pre Operative (Baseline), 1st Assessment (0 Week) and 2nd Assessment (4 week)
  The Borg RPE Scale is a 15-point scale (6 to 20) used to rate subjective experiences during physical exertion. This subjective load scale can help estimate load symptoms, such as the degree of exertion, the degree of load and fatigue.
Length of Hospital stay | Pre Operative (Baseline), 1st Assessment (0 Week) and 2nd Assessment (4 week)
  Total number of days stay in hospital average of days in both group.

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid, MS, Principal Investigator — Riphah International University
Locations (1):
- Rehman Medical Institute, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No